CLINICAL TRIAL: NCT04629859
Title: Malocclusion Patients
Brief Title: Orthognathic Surgeries and Pharyngeal Airway Space
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, principal investigator, Fayoum University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12/10/19
Record Dates: First submitted 2020-11-11; First posted 2020-11-16 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Mandibular Prognathism
Keywords: Orthognathic surgery; Pharyngeal airway space; skeletal class III patients.
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study arm (Experimental): dento skeletal class III patients will undergo a mandibular setback surgery and maxillary advancement
  Interventions: Procedure: mandibular setback and maxillary advancement
- controlled arm (Experimental): dento skeletal class III patients will undergo a mandibular setback surgery
  Interventions: Procedure: mandibular setback

INTERVENTIONS:
Procedure: mandibular setback and maxillary advancement — 12 patients will undergo mandibular setback and maxillary advancement
  Arms: study arm
Procedure: mandibular setback — 12 patients will undergo mandibular setback
  Arms: controlled arm

SUMMARY:
twenty-four patients with dentoskeletal deformity of class III will be divided equally into two groups and will be subjected to orthognathic surgeries group A; will be treated by mandibular setback surgery while group B will be treated with bimaxillary orthognathic surgery in the form of mandibular setback and maxillary advancement surgeries. the total pharyngeal airway will be measured on lateral cephalometric radiographs, integrating retro-palatal and retro-glossal area, and statistically will be compared preoperative, immediate postoperative, and at 6 months post-surgically

ELIGIBILITY:
Inclusion Criteria:

* dento-skeletal class III malocclusion which needed a surgical intervention with maxillary advancement surgery and/or mandibular set-back orthognathic surgery in the form of bilateral sagittal split osteotomy
* no previous orthognathic surgery

Exclusion Criteria:

* Patients with craniofacial syndromes.
* Medically compromised patients and patients with bone anomalies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
total pharyngeal airway space surface area | 6 months
  Cephalometric analyses will be performed, the pharyngeal airway is demarcated inferiorly by a line passing through the tip of epiglottis and the superior tip of the hyoid bone, namely Line A, while the retro-glossal and the retro-palatal airway is separated by a line extending from the basion parallel to line A.
  All the reference points and lines were conveyed to the images . The Pharyngeal airway space was measured and compared.

SECONDARY OUTCOMES:
Epworth sleepiness scale | 6 months
  (0-24) score to assess sleep apnea indirect

CONTACTS AND LOCATIONS:
Overall Officials: hussien hatem, phd, Study Director — Cairo University
Locations (1):
- Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No